CLINICAL TRIAL: NCT00213343
Title: Effects of Phrenic Nerve Stimulation During Swallowing : Experimental Model of Aspiration
Status: Terminated | Type: Observational
Why Stopped: dyspnea
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2002 /149/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Velopharyngeal Insufficiency
Keywords: aspiration; phrenic nerve; magnetic stimulation
MeSH Terms: conditions — Velopharyngeal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
the purpose of this study is to compare the oesophageal depression induced by bilateral phrenic nerve stimulation during swallowing in patients with neurological laryngeal aspiration

DETAILED DESCRIPTION:
phrenic nerve stimulation during swallowing

ELIGIBILITY:
Inclusion Criteria:

stroke with aspiration

Exclusion Criteria:

obstructive rhinitis bronchial obstruction pace maker phrenic nerve paralysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2005-06 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: eric verin, MD -PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France